CLINICAL TRIAL: NCT05002608
Title: A Virtual Health Insurance Navigation for Colorectal Survivors
Brief Title: Virtual Health Insurance Navigation Pilot Program for Colorectal Survivors
Acronym: HINT-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Elyse Park, PhD, Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MGH HINT Colorectal (HINT-C)
Record Dates: First submitted 2021-08-09; First posted 2021-08-12 (Actual); Results first posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Health Insurance; Colorectal Cancer Survivors
Keywords: survivorship

STUDY DESIGN:
Intervention Model Description: Intervention and Usual care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Navigation Intervention (Experimental): The intervention will be delivered via synchronous videoconferencing (real-time delivery and communication between the navigator and the participant) by a trained patient navigator and will consist of 5, 30-minute sessions delivered every week. The navigation intervention group will also receive an online or mailed copy of the health insurance resource guide.
  Interventions: Behavioral: Health Insurance Navigation Tools Program
- Enhanced Usual Care (No Intervention): Enhanced usual care will consist of an online or mailed health insurance resource guide.

INTERVENTIONS:
Behavioral: Health Insurance Navigation Tools Program — The program will be delivered via videoconferencing by a navigator over a 3-month period and will consist of 5 sessions. The navigation intervention sessions will be as follows: Session 1- Insurance Plan Basics; Session 2- Your Plan in Relation to Legal Policy; Session 3- Navigating Your Own Plan and Overcoming Obstacles; Session 4- Managing Care Costs; Session 5- Understanding Your Medical Bills.
  Arms: Navigation Intervention

SUMMARY:
This trial aims to assess the feasibility and acceptability of colorectal survivors approached and engaged in HINT and aims to assess the preliminary efficacy of HINT to improve 1) health insurance literacy and 2) financial burden related to medical cost concerns colorectal survivors. The study investigators propose that, compared to the control arm (who will receive a health insurance information guide, but will not receive the navigation intervention), participants in the HINT intervention arm will have improved health insurance literacy and decreased financial distress related to medical costs.

DETAILED DESCRIPTION:
With support from the American Cancer Society, Dr. Park designed a 5-session health insurance navigation treatment program, Health Insurance Navigation Tools (HINT), that is currently being delivered remotely, as a collaboration with the Childhood Cancer Survivor Study. Given the current insurance landscape and the additional insurance burden that adult colorectal cancer survivors face, the present study seeks to conduct a pilot trial with the existing health insurance intervention and adult colorectal cancer survivors seen at MGH Cancer Centers to improve health insurance literacy and decrease financial burden related to medical costs. The present study seeks to develop and pilot a health insurance navigation program with adult colorectal cancer survivors recruited from MGH. Patients diagnosed with colorectal cancer have a higher risk of experiencing financial burden related to health care costs when compared to patients diagnosed with other types of cancer. While many cancer survivors report experiencing financial burden, financial burden is particularly acute among survivors of colorectal cancer. Outcomes of financial burden among colorectal cancer survivors include lower health related quality of life, employment concerns, and delay or lack of engagement in needed surveillance and follow-up care.

Understanding and navigating insurance benefits in the current landscape is crucial for colorectal cancer survivors to obtain and utilize the health care that they need. With this in mind, the study investigators propose to develop and pilot an insurance navigation intervention to examine its feasibility and acceptability among colorectal cancer survivors receiving care at the MGH.

ELIGIBILITY:
Inclusion Criteria:

* patients who are18-65 years of age
* patients who are 1) approximately 6 months to 5 years posttreatment for stages I-III colon or rectal cancer or 2) approximately more than 3 months post-diagnosis for stage IV colon or rectal cancer at the time of screening
* patients who had a medical visit at MGH in the past two years
* patients who have medical insurance
* patients who speak English
* patients who have access to an iPad, computer, smartphone or laptop with WIFI access

Exclusion Criteria:

* patients who are younger than 18 years of age or older than 65 years of age
* patients who are unable to give consent due to psychiatric or cognitive impairment
* patients who lack of access to a smartphone, computer, or tablet with internet access
* patients who do not currently have health insurance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - MGH, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nekhlyudov L, Walker R, Ziebell R, Rabin B, Nutt S, Chubak J. Cancer survivors' experiences with insurance, finances, and employment: results from a multisite study. J Cancer Surviv. 2016 Dec;10(6):1104-1111. doi: 10.1007/s11764-016-0554-3. Epub 2016 Jun 9. PMID 27277896
- [Background] Rice DR, Farooq A, Hyer JM, Paredes AZ, Bae J, Tsilimigras DI, Pawlik TM. Health expenditures and financial burden among patients with major gastrointestinal cancers relative to other common cancers in the United States. Surgery. 2020 Jun;167(6):985-990. doi: 10.1016/j.surg.2020.02.029. Epub 2020 Apr 15. PMID 32305231
- [Background] Blum-Barnett E, Madrid S, Burnett-Hartman A, Mueller SR, McMullen CK, Dwyer A, Feigelson HS. Financial burden and quality of life among early-onset colorectal cancer survivors: A qualitative analysis. Health Expect. 2019 Oct;22(5):1050-1057. doi: 10.1111/hex.12919. Epub 2019 Jul 5. PMID 31273909
- [Background] Sharp L, O'Leary E, O'Ceilleachair A, Skally M, Hanly P. Financial Impact of Colorectal Cancer and Its Consequences: Associations Between Cancer-Related Financial Stress and Strain and Health-Related Quality of Life. Dis Colon Rectum. 2018 Jan;61(1):27-35. doi: 10.1097/DCR.0000000000000923. PMID 29219919
- [Background] Kent EE, Forsythe LP, Yabroff KR, Weaver KE, de Moor JS, Rodriguez JL, Rowland JH. Are survivors who report cancer-related financial problems more likely to forgo or delay medical care? Cancer. 2013 Oct 15;119(20):3710-7. doi: 10.1002/cncr.28262. Epub 2013 Jul 31. PMID 23907958
- [Background] Ford ME, Sterba KR, Armeson K, Malek AM, Knight KD, Zapka J. Factors Influencing Adherence to Recommended Colorectal Cancer Surveillance: Experiences and Behaviors of Colorectal Cancer Survivors. J Cancer Educ. 2019 Oct;34(5):938-949. doi: 10.1007/s13187-018-1398-5. PMID 30073494
- [Background] Leon AC, Davis LL, Kraemer HC. The role and interpretation of pilot studies in clinical research. J Psychiatr Res. 2011 May;45(5):626-9. doi: 10.1016/j.jpsychires.2010.10.008. Epub 2010 Oct 28. PMID 21035130

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Navigation Intervention | Enhanced Usual Care
Started | 17 | 19
Completed | 15 | 18
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Navigation Intervention | Enhanced Usual Care | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 19 | 36
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (9.5) | 52.6 (7.5) | 52.14 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 9 | 8 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Asian/Pacific Islander | 2 | 1 | 3
  Race/Ethnicity: Black | 0 | 0 | 0
  Race/Ethnicity: Hispanic | 1 | 0 | 1
  Race/Ethnicity: Non-Hispanic White | 14 | 18 | 32
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 19 | 36

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of the Health Insurance Navigation Program
Description: 10-point (1-10; 1= least helpful and 10= most helpful) scale rating of program quality, including the following (higher scores indicate higher levels of acceptability)-
Time Frame: 5 month follow-up
Population: The EUC did not participate in the health insurance navigation so data for this measure was not collected from the EUC arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Navigation Intervention
Number analyzed (Participants) | 15
units on a scale | 8.8 (1.9)

2. Primary Outcome: Change From Baseline Health Insurance Literacy to 5-month Follow-up
Description: 16 items with a 4-category Likert scale ranging from 16-64 (higher scores denoting lower literacy) of confidence on understanding of health insurance terms (higher scores indicate higher levels of health insurance literacy). We report mean health insurance literacy change from baseline to follow-up. Scale adapted from the Urban Institute Health Reform Monitoring Survey-
  * premium
  * deductible
  * co-payments
  * co-insurance
Time Frame: baseline and 5 month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Navigation Intervention | Enhanced Usual Care
Number analyzed (Participants) | 17 | 19
score on a scale | 5.6 (7.5) | 1.1 (9.2)

3. Primary Outcome: Program Feasibility
Description: Program feasibility is measured by the percentage of navigator participants completing all 5 intervention sessions.
Time Frame: 5-month follow-up
Population: The EUC did not complete sessions so data for this measure was not collected from the EUC arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Navigation Intervention
Number analyzed (Participants) | 17
Participants | 15

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Navigation Intervention | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/19
Other Adverse Events (participants affected / at risk) | 0/17 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-29): https://cdn.clinicaltrials.gov/large-docs/08/NCT05002608/Prot_SAP_000.pdf